CLINICAL TRIAL: NCT05108324
Title: Reliability of All on Four Using 2 Zygomatic and 2 Conventional Implants Versus Conventional All on Four Implants Simultaneously for the Rehabilitation of the Atrophied Maxilla (A Randomized Control Trial)
Brief Title: Reliability of All on 4 Using 2 Zygomatic and 2 Conventional Implants vs All on 4 Implants for Rehabilitation of Maxilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mostafa elmasry, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10/11/2021
Record Dates: First submitted 2021-10-11; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Edentulous; Alveolar Process, Atrophy
Keywords: all on four; zygomatic implant
MeSH Terms: conditions — Mouth, Edentulous; Atrophy | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial - parallel group with the patients. It is a superiority trial.
  study group are 10 patients receiving 2 zygomatic implants with 2 conventional implant in anterior region, while the control group are another 10 patients receiving 4 conventional implant 2 in anterior region and 2 in posterior region with immediate loading.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zygomatic implant (Experimental): patients receiving 2 zygomatic implants with 2 conventional implant in anterior region
  Interventions: Procedure: zygomatic implant
- conventional implant (Active Comparator): patients receiving 4 conventional implant 2 in anterior region and 2 in posterior region with immediate loading
  Interventions: Procedure: conventional implant

INTERVENTIONS:
Procedure: zygomatic implant — 2 zygomatic implants and 2 anterior conventional implant
  Other Names: extramaxillary implant
  Arms: zygomatic implant
Procedure: conventional implant — patients will receive 4 conventional dental implant
  Other Names: all on 4
  Arms: conventional implant

SUMMARY:
Oral rehabilitation by dental implants in the severely atrophic maxilla often represents a challenge. To overcome this difficulty, bone augmentation procedures such as sinus augmentation, guided bone regeneration (GBR), or distraction osteogenesis have been used to obtain adequate bone height and width for proper three-dimensional implant placement. To avoid surgical morbidity and shorten treatment length, alternative methods such as short or tilted implants, as well as zygomatic implants (ZIs),have been proposed and have shown promising outcomes.

DETAILED DESCRIPTION:
Placement of dental implants in the pterygo-maxillary region provides adequate posterior bone support for the prosthesis which permits better distribution of masticatory forces without the need of sinus floor augmentation, onlay and inlay grafts, split crest technique, or osteogenic distraction. This allows rehabilitating patients with satisfactory full arch fixed maxillary prosthesis, which is usually spanned from second molar to contralateral second molar tooth.

The purpose of the present study is to compare the Reliability of all on four by 2 zygomatic implants with 2 conventional implant in anterior region versus all on four approach by conventional implant for the rehabilitation of the atrophied maxilla in terms of survival rates and improving the quality of patient's life and involved complication with maxillary sinus.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severely atrophic edentulous upper arch (Cawood class IV, V, VI) that could not be restored with other type of treatment.
2. Patients who had at least 8-12 mm vertical bone height in anterior maxilla to allow installation of at least 2 conventional implants.

Exclusion Criteria:

1. Patients with any systemic disease that might interfere with dental implants placement and/or osseointegration e.g. uncontrolled diabetes, hypertension and osteoporosis, etc.
2. Heavy smoker (> 20 cigarettes daily) and patients with history para-functional habits (e.g. clenching or bruxism, etc.) were also excluded.
3. Intraoral pathological lesion, related to maxilla, maxillary sinus and zygoma.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-10 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-02-14 (Estimated)

PRIMARY OUTCOMES:
change of function of the masticatory muscles | baseline & 6 month after the delivery of the prothesis
  measuring muscles activtiy of masseter and temporalis muscles by electromyography

SECONDARY OUTCOMES:
Implant primary stability | baseline Immediate after implantation
  The implant initial stability will be directly measured after implant insertion using the resonance frequency analysis technique by osttel device

OTHER OUTCOMES:
Biologic complication and implant survival rate | baseline and sixth months
  Any biological complication as sinusitis, fenestration, orbital insults, failure of the implant, are going to be assessed radiographically by the CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed a. Atef, professor, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
data to be shared after publication of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after puplication
Access Criteria: data will be share upon request from Colleges